CLINICAL TRIAL: NCT01288001
Title: A Pilot, Open, Randomised, Controlled, add-on Study Evaluating the Duration of Efficacy of One Intra Articular Injection of Sodium Hyaluronate 2.0% in Patients With Painful Osteoarthritis of the Knee
Brief Title: Study of Evaluating the Duration of Efficacy of One Intra Articular Injection of Sodium Hyaluronate 2.0% in Patients With Painful Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TRB Chemedica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSTP-THA-10-01
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Osteoarthritis Patient

ARMS (1):
- Ostenil plus (Experimental): Patient will get Ostenil plus injection and standard treatment of Osteoarthritis
  Interventions: Drug: Ostenil plus

INTERVENTIONS:
Drug: Ostenil plus — 2% Sodium Hyaluronate plus Mannitol injection

SUMMARY:
A pilot, open, randomised, controlled, add-on study evaluating the duration of efficacy of one intra articular injection of sodium hyaluronate 2.0% in patients with painful osteoarthritis of the knee

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders between 40 and 70 years of age;
2. Primary tibiofemoral osteoarthritis of the knee according to American College of Rheumatology criteria;
3. Pain ≥ 4 on a 10 point scale for at least two out of five subscores of the WOMAC Section A at baseline;
4. Radiologically ascertained grade II or III severity knee osteoarthritis on the Kellgren-Lawrence scale;
5. Having given signed informed consent.

Exclusion Criteria:

1. Secondary knee osteoarthritis, including:

   * septic arthritis;
   * inflammatory joint disease;
   * gout;
   * recurrent episodes of pseudogout;
   * Paget's disease of bone;
   * articular fracture;
   * ochronosis;
   * acromegaly;
   * haemochromatosis;
   * Wilson's disease;
   * primary osteochondromatosis.
2. Clinical signs of acute flare (pain, warm, erythema, effusion of signal knee) at baseline;
3. Axial deviation > 15 degrees in valgus or varus on a standing X-ray;
4. Clinically significant medio-lateral or antero-posterior instability;
5. Rapid destructive arthritis, evolving arthritis requiring surgery within the coming year;
6. Significant injury to the signal knee within 6 months prior to baseline;
7. Complete loss of range of motion;
8. Painful knee conditions other than osteoarthritis (e.g., Sudeck's atrophy, intra-articular neoplasm, villonodular synovitis);
9. Necrosis of one of the femur condyles;
10. History or evidence of gout, chondrocalcinosis;
11. Peripheral neuropathy;
12. Concomitant rheumatic disease:

    * fibromyalgia;
    * rheumatoid arthritis;
    * collagen diseases;
    * psoriatic arthritis and other seronegative spondylarthropathies (e.g., ankylosing spondylitis);
    * metabolic and crystal-induced arthropathies;
    * other osteopathies.
13. Contraindications to intra-articular injection according to investigator's judgement (e.g., local infection at injection site, generalised infection with possible bacteraemia);
14. Skin disease in the area of injection;
15. Severe coagulopathy, ongoing anticoagulation therapy;
16. Accompanying OA of the hip of sufficient severity to interfere with the assessment of the signal knee;
17. Disease of spine, hip or other lower extremity joints of sufficient degree to affect assessment of the signal knee;
18. Poor general health interfering with compliance or assessment;
19. Concomitant disease/ailment other than knee OA requiring the regular use of the patient's normal analgesic medicine;
20. Initiation of chronic treatment with antihistaminics, glucocorticoids, antidepressants or tranquilisers, within less than 3 months prior to baseline;
21. Use of assistive devices other than a cane (walking stick);
22. Surgery of the signal knee other than arthroscopy;
23. Arthroscopy of the signal knee within one year prior to baseline;
24. Treatment with symptomatic slow acting drug for OA (SYSADOA, i.e., chondroitin sulfate, diacerein, glucosamine, piascledine), unless the patient has been on a stable dose for at least 4 months prior to baseline;
25. Intra-articular depocorticosteroid injection into the signal knee within 3 months prior to baseline;
26. Intra-articular SH injection into the signal knee within 6 months prior to baseline;
27. Ascertained hypersensitivity to any product used in the study (SH, paracetamol, diclofenac, omeprazole) or to similar compounds;
28. Pregnant or lactating female;
29. Female of childbearing potential without adequate contraceptive methods;
30. Participation in a drug clinical trial within 3 months prior screening;
31. Patients who, in the judgement of the investigator, will not comply with the protocol.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
to evaluate the duration of efficacy of one intra articular injection of Ostenil® Plus in patients with painful osteoarthritis of the knee. | 6 months
  WOMAC score

SECONDARY OUTCOMES:
to evaluate the effects of the study treatment on pain, joint stiffness, joint function and need for analgesic consumption. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand